CLINICAL TRIAL: NCT02966392
Title: A Randomised Controlled Trial of Continuous Endotracheal Cuff Pressure Control for the Prevention of Ventilator Associated Respiratory Infections
Brief Title: Continuous Endotracheal Cuff Pressure Control to Prevent Ventilator Associated Respiratory Infections
Acronym: VARI-prevent
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oxford University Clinical Research Unit, Vietnam (Other)
Collaborators: The Hospital for Tropical Diseases, Ho Chi Minh City, Vietnam (Unknown); Trung Vuong Hospital, Ho Chi Minh City, Vietnam (Unknown); The National Hospital for Tropical Diseases, Ha Noi, Vietnam (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 16HN
Record Dates: First submitted 2016-11-09; First posted 2016-11-17 (Estimated); Last update posted 2020-05-29 (Actual); Status verified 2020-05

CONDITIONS: Mechanical Ventilation Complication; Tracheal Intubation Morbidity; Ventilator-Associated Pneumonia; Hospital Acquired Infection
Keywords: Cuff pressure; Ventilator associated pneumonia; Respiratory tract infections
MeSH Terms: conditions — Pneumonia, Ventilator-Associated; Cross Infection; Respiratory Tract Infections

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Continuous Pressure Control (CPC) (Experimental): Continuous endotracheal cuff pressure control using Tracoe cuff pressure controller during their intubated stay on ICU.
  Interventions: Device: Tracoe cuff pressure controller
- Standard Care (No Intervention): Intermittent cuff pressure control through manual measurement performed 3 times per day (standard care)

INTERVENTIONS:
Device: Tracoe cuff pressure controller — Participant will be attached to the cuff pressure controller as soon as possible after enrolment. They will remain attached during their intubated stay. If reintubated during same admission they will continue in the intervention arm. If readmitted to ICU they will be managed according to standard care.
  Arms: Continuous Pressure Control (CPC)

SUMMARY:
The purpose of the study is to determine whether automated cuff pressure control results in a reduction in the proportion of patients developing ventilator associated respiratory infections during their stay in intensive care.

DETAILED DESCRIPTION:
The proposed study is a randomized controlled trial of tracheal cuff pressure control using continuous control via an automated electronic device as compared with intermittent pressure control for the prevention of ventilator associated respiratory infection in ICU.

The study will be conducted at multiple sites in Vietnam. Recruitment will be for 18 months at all centers. Patients experiencing any hospital acquired infection whilst at risk of Ventilator Associated Respiratory Infections will be evaluated in using a standardised investigation protocol to identify cases of VARI and other hospital acquired infections (HAI)s. Assessment of VARI will be based on published criteria and carried out by an endpoint review committee independent of patient care and blinded to the allocation of the patient. Antibiotic use data and duration of stay will be important secondary outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* About to be intubated or intubated for ≤ 24 hours (either oral or tracheostomy)
* For active treatment

Exclusion Criteria:

* previously enrolled in this study
* previously intubated within 14 days
* suffering from known tracheomalacia, tracheal stenosis or stridor relating to tracheal injury

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2019-03-07 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
Ventilator Associated Respiratory Infection (VARI) - defined as Ventilator Associated Pneumonia (VAP) or Ventilator Associated Tracheobronchitis (VAT) | From randomisation to ICU discharge/death/transfer or 90 days

SECONDARY OUTCOMES:
Microbiologically confirmed VARI defined as above plus bacterial growth of ≥105 cfu/ml (ETA) or equivalent semi-quantitative for both VAP and VAT | From randomisation to ICU discharge/death/transfer or 90 days
Clinical and microbiologically confirmed VAP (see above for definitions) | From randomisation to ICU discharge/death/transfer or 90 days
Intubated days receiving antibiotics | From randomisation to ICU discharge/death/transfer or 90 days
Incidence of hospital acquired infection | From randomisation to extubation/death/transfer/discharge/ from ICU or 90 days
Total number of days ventilated/in ICU | From randomisation to ICU discharge, death, transfer or 90 days
Cost of ICU stay | From ICU admission to ICU discharge, death, transfer or 90 days
Cost of antibiotics in ICU stay | From ICU admission to ICU discharge, death, transfer or 90 days
Cost of hospital stay | From hospital admission to hospital discharge or 90 days
28 day mortality | From randomisation to 28 days after randomisation
90 day mortality | From randomisation to 90 days after randomisation
ICU mortality | From randomisation to discharge from ICU or death/palliative discharge from it or 90 days
Hospital mortality | From randomisation to discharge from ICU or death/palliative discharge from it or 90 days

OTHER OUTCOMES:
Grade 3 &4 adverse events relating to endotracheal cuff pressure | From randomisation to 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Behzad Nadjm, MBChB MD, Principal Investigator — Oxford University Clinical Research Unit
Locations (3):
- Vietnam (3):
  - National Hospital for Tropical Diseases, Hanoi
  - Hospital for Tropical Diseases, Ho Chi Minh City
  - Trung Vuong Hospital, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: Undecided
We hope to share IPD, however the framework to do so is not yet finalised with our collaborating institutions

REFERENCES:
- [Derived] Dat VQ, Minh Yen L, Thi Loan H, Dinh Phu V, Thien Binh N, Geskus RB, Khanh Trinh DH, Hoang Mai NT, Hoan Phu N, Huong Lan NP, Phuong Thuy T, Vu Trung N, Trung Cap N, Tuyet Trinh D, Thi Hoa N, Thi Thu Van N, Luan VTT, Quynh Nhu TT, Bao Long H, Thanh Ha NT, Thi Thanh Van N, Campbell J, Ahmadnia E, Kestelyn E, Wyncoll D, Thwaites GE, Van Hao N, Chien LT, Van Kinh N, Vinh Chau NV, van Doorn HR, Thwaites CL, Nadjm B. Effectiveness of Continuous Endotracheal Cuff Pressure Control for the Prevention of Ventilator-Associated Respiratory Infections: An Open-Label Randomized, Controlled Trial. Clin Infect Dis. 2022 May 30;74(10):1795-1803. doi: 10.1093/cid/ciab724. PMID 34420048
- [Derived] Dat VQ, Geskus RB, Wolbers M, Loan HT, Yen LM, Binh NT, Chien LT, Mai NTH, Phu NH, Lan NPH, Hao NV, Long HB, Thuy TP, Kinh NV, Trung NV, Phu VD, Cap NT, Trinh DT, Campbell J, Kestelyn E, Wertheim HFL, Wyncoll D, Thwaites GE, van Doorn HR, Thwaites CL, Nadjm B. Continuous versus intermittent endotracheal cuff pressure control for the prevention of ventilator-associated respiratory infections in Vietnam: study protocol for a randomised controlled trial. Trials. 2018 Apr 4;19(1):217. doi: 10.1186/s13063-018-2587-6. PMID 29615093